CLINICAL TRIAL: NCT02029807
Title: Comparison of Compensatory Reserve Index to Intravascular Volume Change and Stroke Volume During Blood Donation
Brief Title: Comparison of Physiological Variables During Blood Donation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Flashback Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-2334
Record Dates: First submitted 2013-12-16; First posted 2014-01-08 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood donors: Healthy adult volunteers donating blood

SUMMARY:
The investigators have developed a system based on a pulse oximeter, a tablet, and an algorithm running on the tablet that analyzes the pulse oximeter waveform.

The algorithm that runs on this system should be able to accurately keep track of blood loss during blood donation. The investigators will compare the algorithm with the blood loss tracked by a device called a flow meter.

The algorithm that runs on this system should be able to accurately keep track of stroke volume changes. The investigators will compare the algorithm with the stroke volume changes tracked by a device called a CCNexfin.

The algorithm that runs on this system should work whether it's in place for the whole blood donation, or if it's placed after the blood donation has started. The investigators will use two pulse oximeters for the system on each hand and compare one that is used for the whole blood donation versus one that is not used for the whole blood donation.

DETAILED DESCRIPTION:
Hypothesis: p-values for testing the hypothesis of no correlation against the alternative that there is a nonzero correlation for each subject will be calculated. The minimum average power correlation, alpha = 0.05, will be used. Correlation will be made (CRI trend during 550ml blood volume removal) using pre and post blood draw data.

Specific Aims: These data will be submitted to the FDA with the following claims: The CRI algorithm

1. Is intended for use by clinicians and medically qualified personnel to noninvasively display the trend of intravascular volume changes (hemorrhage)
2. Is intended for use by clinicians and medically qualified personnel to noninvasively display the trend of stroke volume changes and
3. The CRI trend value is not relative to an initial CRI reading, instead it is an actual CRI trend value that does

ELIGIBILITY:
Inclusion Criteria:

* Subject is planning on donating blood and is approved by Children's Hospital Colorado's Blood Donation Center
* Age 18-89 years
* Previously donated blood (lower likelihood of vasovagal response)

Exclusion Criteria:

* Pregnant
* Incarcerated
* Limited access to or compromised monitoring sites for non-invasive finger sensors

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers donating blood
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Intravascular volume | Day One
  The CRI algorithm is intended to display the trend of intravascular volume changes. This is measured Day One.
Change in Stroke volume | Day One
  The CRI algorithm is intended to display the trend of stroke volume changes. This is measured Day One.
CRI trend | Day One
  The CRI algorithm is intended to not require calibration, or being placed, during normal physiological conditions. This is measured Day One.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado's Blood Donation Center, Aurora, Colorado, United States